CLINICAL TRIAL: NCT02818634
Title: Effect of Costal Harvesting Technique on Postoperative Donor-site Morbidity: Does Muscle Sparing Technique Cause Less Postoperative Pain ? A Clinical Trial
Acronym: COSTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Berke Ozucer, MD, Otolaryngologist, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COSTA
Record Dates: First submitted 2016-06-17; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Nasal Deformity; Revision Rhinoplasty; Autogenous Rib Graft; Costal Cartilage; Harvesting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Muscle-sparing (Active Comparator): Following skin incision with No.15 blade; all layers including the subcutaneous fat, muscle fascia and muscles covering the cartilage were passed with blunt dissection. Muscle fibers were dissected parallel to their positioning.
  Interventions: Procedure: Harvesting rib cartilage
- Muscle-cutting (Active Comparator): Following skin incision with No.15 blade; all layers including the subcutaneous fat, muscle fascia and muscles covering the cartilage were cut with Monopolar electrocautery at (25 watts).
  Interventions: Procedure: Harvesting rib cartilage

INTERVENTIONS:
Procedure: Harvesting rib cartilage

SUMMARY:
The purpose of this study was to investigate the effect of 'muscle sparing technique' while harvesting costal/rib cartilage on postoperative donor-site morbidity -namely postoperative pain. Although authors report 'muscle sparing technique' cause less pain its not investigated in an evidence-based-medicine perspective. Therefore the investigators are planning a controlled, prospective clinical trial to compare the conventional method and 'muscle sparing technique'.

Effect of Costal Harvesting Technique on Postoperative Donor-site Morbidity: Does Muscle Sparing Technique Cause Less Postoperative Pain ? A Clinical Trial

DETAILED DESCRIPTION:
Revision rhinoplasty patients requiring costal cartilage were enrolled in the study. All costal cartilage harvestings were full-thickness and they were carried out by a single-surgeon (Berke Ozucer). Patients were randomly assigned either to 'Conservative Muscle-cuttingHarvesting Technique' or 'Muscle-sparing Harvesting Technique'.

Surgical technique costal cartilage harvesting in both groups were identical expect this:

M-Cutting group : Following skin incision with No.15 blade; all layers including the subcutaneous fat, muscle fascia and muscles covering the cartilage were cut with Monopolar electrocautery at (25 watts).

M-Sparing group: : Following skin incision with No.15 blade; all layers including the subcutaneous fat, muscle fascia and muscles covering the cartilage were passed with blunt dissection. Muscle fibers were dissected parallel to their positioning.

Postoperative pain was evaluated with a Visual Analogue Scale. Participants were questioned regarding their donor-site pain and asked to score their pain 0 (minimum and 10 (maximum). Passive state and pain while active was evaluated separately. This evaluation was carried out at 6th postoperative hour, first, second, third postoperative-days, first postoperative week, on 15th ,30th and 45th day postoperatively. Also postoperative need for analgesics were also noted for the first three days.

Muscle-cutting and muscle-sparing groups were analysed for mean ± Standard deviation values. These values were compared statistically to assess whether muscle-sparing technique has a significant effect on reduced postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Revision rhinoplasty
* when costal cartilage is harvested full-thickness

Exclusion Criteria:

* Fibromyalgia
* No consent
* When patient does not comply with follow-up

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in Postoperative Pain | Postoperative first 45 days
  Postoperative pain and its change from baseline to 45th postoperative day will be evaluated with Visual Analogue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Berke Ozucer, MD, Study Director — Gaziosmanpasa Taksim Research and Education Hospital, Otorhinolaryngology Deparment; Mehmet E Dinc, MD, Principal Investigator — Gaziosmanpasa Taksim Research and Education Hospital, Otorhinolaryngology Deparment
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Department of Otorhinolaryngology, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

REFERENCES:
- [Background] Fedok FG. Costal Cartilage Grafts in Rhinoplasty. Clin Plast Surg. 2016 Jan;43(1):201-12. doi: 10.1016/j.cps.2015.08.002. Epub 2015 Oct 24. PMID 26616708
- [Background] Cochran CS. Harvesting Rib Cartilage in Primary and Secondary Rhinoplasty. Clin Plast Surg. 2016 Jan;43(1):195-200. doi: 10.1016/j.cps.2015.09.018. Epub 2015 Oct 23. PMID 26616707